CLINICAL TRIAL: NCT03551964
Title: Cangrelor Versus Ticagrelor In Patients With Acute Myocardial Infarction Complicated With Initial Cardiogenic Shock
Brief Title: Dual Antiplatelet Therapy For Shock Patients With Acute Myocardial Infarction
Acronym: DAPT-SHOCK-AMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Collaborators: Charles University, Czech Republic (Other); Masaryk University (Other); Ministry of Health, Czech Republic (Other Government); National Institute for Metabolic and Cardiovascular Disease Research (Unknown); Institute of Hematology and Blood Transfusion, Czech Republic (Other); BioVendor LM (Unknown)
Responsible Party: Principal Investigator, Zuzana Motovska, Zuzana Motovska MD PHD, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13062017-23-1; 2018-002161-19 (EudraCT Number)
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Acute Myocardial Infarction; Cardiogenic Shock
Keywords: Acute myocardial infarction; Cardiogenic shock; Primary percutaneous coronary intervention; Dual antiplatelet therapy; Cangrelor; Ticagrelor
MeSH Terms: conditions — Shock, Cardiogenic | interventions — cangrelor; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cangrelor therapy (Experimental): IV Cangrelor is initiated immediately after the patient arrives at the 24/7 PCI center (cathlab, coronary/intensive care unit, other parts of department) and is randomized to the study.
  Interventions: Drug: Cangrelor
- Ticagrelor therapy (Active Comparator): The patient will receive the initial dose of crushed Ticagrelor immediately after arriving at the 24/7 PCI center (cath lab, coronary/intensive care unit, other parts of the department) and after being randomly assigned to the study; in patients with a disorder of consciousness, the initial dose will be administered immediately after the nasogastric tube is inserted.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Cangrelor — Cangrelor: IV bolus 30 µg/kg (application < 1 minute) followed immediately by continuous infusion at 4 µg/kg. Tables to calculate bolus dose in ml and infusion (in ml per hour) rate for each body weight group will be prepared in advance and will be included in the study medication kit to accelerate treatment start.
  * Cangrelor treatment will be discontinued after circulatory stabilization (but no earlier than 2 hours after infusion initiation) i.e. after systolic Blood Pressure (sBP) is maintained at the level > 100 mmHg for one hour after the end of IABK and/or vasoactive treatment is discontinued, but no later than 4 hours after PCI,
  * 30 minutes before the end of Cangrelor infusion, administration of Ticagrelor 180 mg (crushed tablets) and then dose 90 mg every 12 hours.
  Other Names: intravenous P2Y12 inhibitor
  Arms: Cangrelor therapy
Drug: Ticagrelor — Ticagrelor: 180 mg loading dose - crushed tablets, 2 x 90 mg maintenance dose
  Other Names: oral P2Y12 inhibitor
  Arms: Ticagrelor therapy

SUMMARY:
Multicenter, international, randomized, placebo-controlled, double-blind trial comparing intravenous cangrelor and crushed oral ticagrelor in patients with acute myocardial infarction complicated by initial cardiogenic shock (CS-AMI) and treated with primary angioplasty (PCI).

The Dual Antiplatelet Therapy For Shock Patients With Acute Myocardial Infarction (DAPT-SHOCK-AMI) trial tests the hypothesis that intravenous cangrelor is (a) more effective in terms of its rate of onset and the proportion of patients achieving effective periprocedural inhibition of ADP-induced platelet aggregation and (b) at least as effective as the recommended treatment of oral (crushed) ticagrelor in reducing major cardiovascular events in patients with initial CS-AMI indicated for primary PCI strategy.

DETAILED DESCRIPTION:
Randomization to study drugs will be performed using an online database system for data collection. After entering basic patient data, the assigned arm and the randomization code will be generated based on a predefined randomization scheme.

Concomitant therapy includes acetylsalicylic acid: an initial intravenous dose of 500 mg, followed by a daily oral dose of 100 mg. A proton pump inhibitor is also recommended. Additional therapies, such as further antithrombotic treatments (e.g., GP IIb/IIIa inhibitors, heparin) and mechanical support (IABP, ECMO), remain fully within the competence of the treating physician.

Electronic database - eCRF. The data from individual follow-up assessments will be entered into an electronic database. The online instrument CLADE-IS will be used for data collection; this instrument provides robust options for electronic case report form (eCRF) design, hierarchical administration of user rights and a user-friendly web interface. The system provides predefined validation rules, conversions of variables, and it considers the relationships between variables; user access is controlled by the hierarchical system of user rights and user roles, and database operations are stored for audits and tracking of changes. Data safety is ensured through physical security of the servers, authorized access, and backup procedures.

Laboratory collections. The efficacy of the antiplatelet drugs cangrelor and ticagrelor will be determined using flow cytometry analysis of intracellular VASP (vasodilator-stimulated phosphoprotein) phosphorylation.

Study Committees: Executive c., Steering c., Endpoint adjudication c., Data safety monitoring board.

Monitoring. External monitor Clinical Research Associate (CRA)

Definitions.

Death is defined as death from all causes.

Death from cardiovascular causes is defined as a death with evidence of a cardiovascular cause or any death without clear evidence of a non-cardiovascular cause. All deaths are considered cardiac unless a clear non-cardiac cause can be identified. Any unexpected death (for example, in patients with a co-existing, potentially fatal non-cardiac disease such as cancer or infection) is classified as a death from cardiovascular causes.

Myocardial reinfarction (MI) is defined as a new (additional) MI that must differ from the MI based on which the patient was enrolled into the study, satisfying the universal definition of MI criteria.

Urgent revascularization of the infarct-related artery is defined as a new emergent/urgent revascularization of the artery that was intervened in during the initial procedure due to repeated manifestations of ischemia after the completion of the initial PCI.

Stroke is defined as the rapid onset of a new neurological deficit due to an ischemic or hemorrhagic lesion in the central nervous system, with symptoms lasting at least 24 hours from their onset or resulting in death.

Definitive stent thrombosis is defined according to the Academic Research Consortium criteria.

New heart failure is defined as a hospitalization or emergency check-up for heart failure in a doctor's office or emergency room that requires treatment.

Bleeding is defined according to the Bleeding Academic Research Consortium (BARC) criteria.

External collaborating centre for data-management and statistical analyses: Institute of Biostatistics and Analyses at the Faculty of Medicine of the Masaryk University in Brno, Czech Republic.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Acute myocardial infarction according to the definition of ESC/ACC/AHA, indicated for emergency percutaneous coronary intervention (primary PCI strategy)
3. Cardiogenic shock present upon admission due to the AMI (≥ 2 of the criteria below are satisfied)

   1. sBP < 90 mmHg with the absence of hypovolemia
   2. Need of vasopressor and/or inotropic therapy
   3. Presence of the signs of the organ hypoperfusion - cyanosis, cold acra, disorder of consciousness, congestive heart failure
4. Informed consent form signed
5. Women of childbearing potential should be protected from pregnancy throughout the study (relevant for long-term use of ticagrelor). Suitable methods of contraception in this case include hormonal contraceptives, barrier methods, or complete withdrawal - as long as it is consistent with the patient's lifestyle.

Exclusion Criteria:

1. Contraindications of antiplatelet therapy with ticagrelor/cangrelor

   * Recent (< 6 months) major bleeding
   * Recent (< 1 month) major surgery/injury
   * History of intracranial bleeding
   * History of stroke/TIA
   * Known intolerance to ticagrelor/cangrelor
   * Severe impairment of hepatic function
   * Concomitant administration of strong CYP3A4 inhibitors (for example, ketoconazole, clarithromycin, nefazodone, ritonavir, and atazanavir)
2. Administration of a loading dose of an oral P2Y12 inhibitor prior to admission (clopidogrel ≥ 300 mg, ticagrelor 180 mg, prasugrel 60 mg)
3. Need of concomitant chronic anticoagulation therapy due to indications such as atrial fibrillation, artificial valve, thromboembolic disease, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Primary Laboratory endpoint | At the end of primary percutaneous coronary intervention; Within 24 hours from randomization
  The periprocedural rate of onset and the proportion of patients who achieve effective* P2Y12 platelet receptor inhibition defined by a Platelet Reactivity Index (PRI) value.
  *PRI less than 50% as measured by the vasodilator-stimulated phosphoprotein phosphorylation flow cytometric assay
Primary Clinical Endpoint | Within 30 days after randomization
  The composite of all-cause death, myocardial infarction, or ischemic stroke expressed as a proportion of patients with any of these events.

SECONDARY OUTCOMES:
Key secondary efficacy endpoint | Within 30 days and one year after randomization
  Death, myocardial infarction, urgent revascularization of the infarct-related artery, stent thrombosis, or ischemic stroke expressed as a proportion of patients with any of these events
Key secondary safety endpoint | Within 30 days and one year after randomization
  Bleeding as defined by BARC type ≥ 3B, expressed as a proportion of patients with this event.
Secondary net-clinical endpoint | Within 30 days and one year after randomization
  Death, myocardial infarction, urgent revascularization of the infarct-related artery, stroke, or major bleeding as defined by the BARC type ≥ 3B criteria expressed as a proportion of patients with any of these events.
Secondary efficacy endpoint | Within 30 days and one year after randomization
  Cardiovascular death, myocardial infarction, urgent revascularization, and heart failure expressed as a proportion of patients with any of these events.
Secondary endpoint | Within 30 days and one year after randomization
  Heart failure, expressed as a proportion of patients with this event.
Other secondary outcome | Within 30 days and one year after randomization
  Individual components of the primary clinical endpoint.
Other secondary efficacy endpoint | Within 30 days and one year after randomization
  Death from cardiovascular causes, expressed as a proportion of patients with this event.
Other secondary endpoint | Within 30 days after randomization
  Definite stent thrombosis, expressed as a proportion of patients with this event.
Secondary safety endpoint | Within 30 days after randomization
  Bleeding as defined by BARC type ≥ 3B, expressed as a proportion of patients with this event.
Other secondary outcome | Within 30 days after randomization
  Delayed* aortocoronary bypass surgery due to a risk of bleeding.
  *Assessed by the heart team, indicating aortocoronary bypass surgery.
Secondary laboratory endpoint | 1 hour after primary PCI
  Effective* P2Y12 platelet receptor inhibition defined by Platelet Reactivity Index (PRI) value
  *PRI less than 50% as measured by the vasodilator-stimulated phosphoprotein phosphorylation flow cytometric assay
Secondary endpoint | From randomization to end of index event hospitalization, within 3 months after randomization
  Duration of hospitalization* in days
  *Intensive care unit stay and total hospital stay
Other secondary endpoint | Initial phase of index event hospitalization, within 7 days after randomization
  Maximum values of high-sensitive cardiac troponin in μg per liter
Secondary outcome | From randomization to the end of vasoactive pharmacotherapy / mechanical circulatory support, within 30 days after randomization
  Duration of vasoactive pharmacotherapy and/or mechanical circulatory support in days

OTHER OUTCOMES:
Cost analysis | Within 30 day and one year after randomization
  Cost-effectiveness analysis
MRI sub-study endpoints | Within one year after randomization
  Magnetic Resonance Imaging sub-study
Echo sub-study endpoints | Within one year after randomization
  Echocardiographic substudy

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Motovska, MD, PhD., Principal Investigator — University Hospital Kralovske Vinohrady, Charles University, Prague, Czech Republic; Deepak L Bhatt, MD, MPH, MBA., Principal Investigator — Mount Sinai Fuster Heart Hospital, Icahn School of Medicine at Mount Sinai, New York, NY, USA
Locations (29):
- Czechia (18):
  - University Hospital Kralovske Vinohrady, Prague, Please Select
  - St. Anne's University Hospital Brno, Brno
  - Department of Cardiology, University Hospital Brno-Bohunice, Brno
  - Cardiology Department, Regional Hospital, České Budějovice
  - University Hospital Hradec Králové, Hradec Králové
  - Cardiology department, Regional hospital, Jihlava
  - Cardiocenter, Regional Hospital, Karlovy Vary
  - Krajská nemocnice Liberec, Liberec
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
  - Department of Cardiology, Regional Hospital,, Pardubice
  - University Hospital Pilsen, Pilsen
  - General University Hospital in Prague, Prague
  - Institute of Clinical and Experimental Medicine, Prague
  - Na Homolce Hospital, Prague
  - Cardiocenter, Hospital Podlesi, Třinec
  - Masaryk Hospital, Ústí nad Labem
  - Regional Hospital T. Bati, Zlín
- France (2):
  - Département de Cardiologie, Hôpital Bichat Assistance Publique Hôpitaux de Paris, Paris
  - Pitié-Salpêtrière Hospital (AP-HP), Paris
- Germany (3):
  - Heart Center Freiburg University, Freiburg im Breisgau
  - University Medical Centre, Mannheim
  - University Hospital Tübingen, Tübingen
- Poland (3):
  - Collegium Medicum University Hospital No. 1, Bydgoszcz
  - Jagiellonianan University, University Hospital Krakow, Krakow
  - Medical University of Warsaw, Warsaw
- Slovakia (3):
  - Middle-Slovak Institute of Cardiovascular Diseases, Banská Bystrica
  - Center of Interventional Neuroradiology and Endovascular Treatment, Bratislava
  - Cardiocentre, Nitra

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Motovska Z, Hlinomaz O, Mrozek J, Kala P, Geisler T, Hromadka M, Akin I, Precek J, Kettner J, Cervinka P, Montalescot G, Jarkovsky J, Belohlavek J, Bis J, Matejka J, Vodzinska A, Muzafarova T, Tomasov P, Schee A, Bartus S, Andrasova A, Olivier CB, Kovarik A, Ostadal P, Demlova R, Souckova L, Vulev I, Coufal Z, Kochman J, Marinov I, Kubica J, Ducrocq G, Karpisek M, Klimsa Z, Hudec M, Widimsky P, Bhatt DL, Group DS. Cangrelor versus crushed ticagrelor in patients with acute myocardial infarction and cardiogenic shock: rationale and design of the randomised, double-blind DAPT-SHOCK-AMI trial. EuroIntervention. 2024 Oct 21;20(20):e1309-e1318. doi: 10.4244/EIJ-D-24-00203. PMID 39432252
- [Derived] Filipescu R, Collins SP, Radu RI, Ben Gal T, Antohi L, Abdelhamid M, Geavlete O, Pana M, Farmakis D, Matei DC, Savarese G, Margineanu C, Polovina M, Miro O, Guz D, Palazzuoli A, Masip J, Adamo M, Ambrosy AP, Chioncel O. Therapeutic Advances in the Management of Cardiogenic Shock. Am J Ther. 2026 Jan 15. doi: 10.1097/MJT.0000000000002025. Online ahead of print. PMID 41543923
- [Derived] Connery A, Ahuja T, Katz A, Arnouk S, Zhu E, Papadopoulos J, Rao S, Merchan C. Antithrombotic Stewardship: Evaluation of Platelet Reactivity-Guided Cangrelor Dosing Using the VerifyNow Assay. J Cardiovasc Pharmacol. 2024 May 1;83(5):482-489. doi: 10.1097/FJC.0000000000001543. PMID 38335531

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT03551964/SAP_001.pdf